CLINICAL TRIAL: NCT01045889
Title: First Line Treatment in HIV-related Large Cell Non Hodgkin Lymphoma at "High Risk", Including Early Consolidation With High Dose Chemotherapy and Autologous Peripheral Blood Stem Cell Transplantation
Brief Title: High Dose Therapy and Peripheral Blood Stem Cell Transplantation in HIV Related Non Hodgkin Lymphoma (NHL) at High Risk
Acronym: HDT-HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Giuseppe Rossi, Director of Hematology, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ema2_LNH e HIV
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: HIV-related Lymphoma; HIV Infections
Keywords: HIV; non hodgkin lymphoma; peripheral blood stem cell transplantation
MeSH Terms: conditions — Lymphoma, AIDS-Related; HIV Infections; Lymphoma, Non-Hodgkin | interventions — Rituximab; VAP-cyclo protocol; Peripheral Blood Stem Cell Transplantation; Cyclophosphamide; Vincristine; Prednisone; Carmustine; Etoposide; Cytarabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- R-CHOP + PBSCT (Experimental): All patients will receive chemoimmunotherapy with Rituximab + CHOP regimen for 6 cycles followed by high dose cyclophosphamide and stem cell collection, then high dose therapy with BEAM conditioning regimen and peripheral blood stem cell transplantation
  Interventions: Other: Rituximab and CHOP regimen + PBSCT

INTERVENTIONS:
Other: Rituximab and CHOP regimen + PBSCT
  Other Names: Mabthera; cyclophosphamide; adryamicin; vincristine; prednisone; BiCNU; etoposide; aracytin; melphalan

SUMMARY:
The purpose of the study is to evaluate the efficacy of an intensified first-line treatment, with conventional chemotherapy (CHOP) plus monoclonal antibody anti CD20, followed by high dose chemotherapy and PBSC transplantation in HIV-related aggressive non-Hodgkin lymphoma at "high risk" , according to the international prognostic index (IPI).

DETAILED DESCRIPTION:
HIV associated NHL show particularly aggressive clinical features and a worse prognosis compared to the general population. The recent introduction of highly active antiretroviral therapy (HAART)has improved HIV positive patients' clinical conditions and reduced the risk of opportunistic infections, thus making HIV+ patients more similar to HIV- patients. Several studies have shown that the early use (as first line treatment) of high dose chemotherapy (HDT) with peripheral blood stem cell transplantation (PBSCT) is superior in the HIV negative setting to conventional dose chemotherapy, at least in patients with poor prognostic factors at diagnosis. Recently, several experiences have shown the feasibility, safety and efficacy of HDT and PBSCT, in association with HAART, as salvage therapy in HIV positive patients with lymphoma who maintain a chemosensitive disease after first-line treatment failure. It is rationale therefore to explore the use of this treatment strategy earlier, within the upfront treatment of HIV-associated lymphoma, in those patients with poor prognostic factors at diagnosis, according to the international prognostic score (IPI).

ELIGIBILITY:
Inclusion Criteria:

* HIV positivity
* "Large cell"histology (DLBCL, Immunoblastic, Plasmablastic, Anaplastic lymphoma)
* Age 18-60 years
* Age-adjusted IPI 2-3
* Ann Arbor stage I B-IV
* Written informed consent.

Exclusion Criteria:

* Burkitt lymphoma
* Lymphoblastic lymphoma
* Primary effusion lymphoma
* Age-adjusted IPI 0-1
* Performance Status (WHO) >2 (if not related to lymphoma)
* Inadequate cardiac function (V.E.F. < 50%) or clinically evident cardiac disease
* Inadequate pulmonary function (DLCO < 50% and/or O2 < 96%)
* Inadequate renal function (creatinine > 2 mg/dl)
* Inadequate liver function (AST/ALT > 3 ULN and/or PT < 70%, if not related to lymphoma)
* Inadequate marrow function (neutrophils < 1500/cmm; platelets < 100.000/cmm, if not related to lymphoma)
* Virologic failure to HAART (including at least one NRTI, one NNRTI and two PI) and/or CD4 count < 50/cmm.
* CNS or meningeal lymphoma
* Active opportunistic infections
* Pregnancy
* Other evolutive malignancy (except of localized non-melanoma skin cancer and in situ portio carcinoma)
* Any other condition that contraindicates this treatment program at discretion of physician
* HBsAg positivity with active viral replication (HBV-DNA positivity)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2007-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2-years

SECONDARY OUTCOMES:
Partial and complete responses | Evaluation of response one month after peripheral blood transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Rossi, MD, Principal Investigator — Haematology Division - AO Spedali Civili di Brescia - Italy
Locations (1):
- AO Spedali Civili di Brescia, Brescia, Italy, Italy

REFERENCES:
- [Background] Re A, Michieli M, Casari S, Allione B, Cattaneo C, Rupolo M, Spina M, Manuele R, Vaccher E, Mazzucato M, Abbruzzese L, Ferremi P, Carosi G, Tirelli U, Rossi G. High-dose therapy and autologous peripheral blood stem cell transplantation as salvage treatment for AIDS-related lymphoma: long-term results of the Italian Cooperative Group on AIDS and Tumors (GICAT) study with analysis of prognostic factors. Blood. 2009 Aug 13;114(7):1306-13. doi: 10.1182/blood-2009-02-202762. Epub 2009 May 18. PMID 19451551